CLINICAL TRIAL: NCT03052309
Title: BIOTRONIK - A Prospective, International, Multi-centre, Post-market All-comers Registry to Assess the Clinical Performance of the Passeo-18 Lux Paclitaxel Releasing Balloon Catheter in Popliteal Arteries - III BENELUX
Brief Title: BIOLUX P-III BENELUX All-Comers Registry
Status: Completed | Type: Observational
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Other Study IDs: C1604
Record Dates: First submitted 2017-02-02; First posted 2017-02-14 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Passeo-18 Lux DCB — The decision to treat the patient with Passeo-18 DCB is at the investigator discretion. The endovascular procedure is performed as per standard of care and device Instructions For Use (IFU)

SUMMARY:
The purpose of the BIOLUX P-III BENELUX Registry is to further investigate the safety and clinical performance of the Passeo-18 Lux Drug Coated Ballon when used in daily clinical practice for the treatment of isolated atherosclerotic lesion (vessel narrowing) in popliteal arteries

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or minimum age as required by local regulations
* Subject must be willing to sign a Patient Data Release Form (PDRF) or Patient Informed Consent (PIC) where applicable
* Lesion(s) in the popliteal arteries suitable for endovascular treatment, treated with or scheduled to be treated with the Passeo-18 Lux drug coated balloon.
* Isolated popliteal artery lesion: at least 2 cm of healthy segment between lesion(s) in the popliteal artery and lesion(s) in distal superficial femoral artery
* Inflow free from flow-limiting lesion. Patients with flow-limiting inflow lesions (> 50% stenosis) can be included if lesion(s) have been treated successfully before or during the index procedure, with a maximum residual stenosis of 30% per visual assessment
* At least one native artery with direct outflow artery to the foot
* Rutherford classification 2-5
* Patient with bypass surgery in the same limb can be enrolled if there is at least 2 cm healthy segment between popliteal artery and anastomosis

Exclusion Criteria:

* Life expectancy ≤ 1 year
* Rutherford classification 6
* Lesion involving the superficial femoral artery (arterial intersection with the femur in an anteroposterior view) or extending in infra-popliteal arteries (origin of the anterior tibial artery or tibioperoneal trunk)
* Aneurysm at the level of the popliteal artery
* Failure to successfully cross the target lesion with a guide wire (successful crossing means tip of the guide wire distal to the target lesion in the absence of flow limiting dissections or perforations)
* Intraprocedural decision not to proceed with the Passeo18 Lux DCB for any reason not related to the device (for instance blood flow limiting dissection after predilatation)
* Subject is currently participating in another investigational drug or device study that has not reached its primary endpoint yet
* Subject is pregnant or planning to become pregnant during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The BIOLUX P-III BENELUX registry will include subjects from an all-comers patient population with all subjects requiring popliteal artery revascularization with the Passeo-18 Lux DCB
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Freedom from Major Adverse Events (MAE) | 6 months
  Freedom from Major Adverse Events (MAE): A composite of freedom from device- and procedure-related mortality through 30 days, and freedom from major target limb amputation and clinically driven target lesion revascularization (TLR)
Freedom from clinically driven target lesion revascularization (cd-TLR) | 12 months
  Any re-intervention performed for ≥ 50% diameter stenosis (visual estimate) at the target lesion after documentation of recurrent clinical symptoms of the patient.)

SECONDARY OUTCOMES:
Freedom from clinically-driven target lesion revascularization (cd-TLR) | 6 and 24 months
Freedom from clinically-driven target vessel revascularization (TVR) | 6, 12 and 24 months
Primary patency | 12 and 24 months
  freedom from >50% restenosis in the target lesion as indicated by a duplex ultrasound peak systolic velocity ratio (PSVR) >2.5 or by visual assessment of an angiogram with no clinically driven re-intervention
Freedom from Major Adverse Events (MAE) | 12 and 24 months
  Freedom from Major Adverse Events (MAE): A composite of freedom from device- and procedure-related mortality through 30 days, and freedom from major target limb amputation and clinically driven target lesion revascularization (TLR)
Change in mean Ankle Brachial Index (ABI) | 6, 12 and 24 months
  compared to the pre-procedure
Improvement in Rutherford classification | 6, 12 and 24 months
  compared to the pre-procedure Rutherford classification
Amputation-free survival (AFS) | 6, 12 and 24 months
  including major, minor and overall AFS
Pain score | 6, 12 and 24 months
  compared to the pre-procedure score.
Walking Impairment Questionnaire | 6, 12 and 24 months
  compared to the pre-procedure score.
Device success | immediately upon index procedure
  Successful delivery, inflation, deflation, and retrieval of the Passeo-18 Lux DCB
Technical success | immediately upon index procedure
  Successful completion of the endovascular procedure and immediate morphological success with ≤ 50% residual diameter reduction of the treated lesion as determined by visual estimation
Procedural success | immediately upon discharge
  Procedural success is technical and device success without the occurrence of any MAE (as defined in the protocol) during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Franck Vermassen, Principal Investigator — UZ Gent; JGAM Blomjous, Principal Investigator — OLVG Amsterdam
Locations (9):
- Belgium (5):
  - Ziekenhuis Oost Limburg Genk, Genk
  - University Hospital Gent (UZ Gent), Ghent
  - Algemeen Ziekenhuis Groeninge Kortrijk, Kortrijk
  - Algemeen Ziekenhuis Delta Roeselare, Roeselare
  - AZ Portaels, Vilvoorde
- Centre Hospitaliers Luxembourg, Luxembourg, Luxembourg
- Netherlands (3):
  - OLVG, Amsterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Maxima Medisch Centrum Veldhoven, Veldhoven

IPD SHARING:
Plan to Share IPD: No